CLINICAL TRIAL: NCT06547723
Title: Developing and Compiling a Mindfulness-Based Stress Reduction Program and Evaluating Its Effectiveness on Relieving Chronic Pain in the Elderly
Brief Title: MBSR Program and Evaluating Its Effectiveness on Relieving Chronic Pain in the Elderly
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Soukhtanlou (Other)
Responsible Party: Sponsor-Investigator, Mohammad Soukhtanlou, Mohammad Soukhtanlou M.Sc., University of Tehran
Organization: University of Tehran (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UTehran
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
Keywords: Mindfulness-based stress reduction program; Chronic pain; Elderly; Physiotherapy
MeSH Terms: conditions — Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This is a feasibility study with a control group along with randomized double-blind parallel groups on 40 elderly patients with chronic pain.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, simple individual randomization method is used. None of the participants and researchers will be informed about the placement of the participants in the groups until the start of the project, and for this purpose, spss software will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Participants in the experimental group receive 20 sessions physiotherapy (in first-4-week, three sessions and next-4-week two sessions on a weekly basis) along with one MBSR session (total MBSR sessions are eight sessions), which also include regular MBSR homework.
  Interventions: Other: MBSR and physiotherapy
- control group (Active Comparator): Participants in the control group receive 20 sessions physiotherapy (in first-4-week, three sessions and next-4-week two sessions on a weekly basis).
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: MBSR and physiotherapy — In experimental group in the first session, the research program and plans for outcome assessment will be introduced. They will sign the research agreement form and will be interviewed to obtain information about their pain, their medication(s), and demographics. This will be followed by the first 70-80-minute physiotherapy session. During each session, the physiotherapist will administer the Transcutaneous electrical nerve stimulation (TENS), low-level laser therapy (LLLT), and ultrasound therapy to the painful body region. In addition, they will engage in 20 minutes of exercise during each session.
  After that, participants will be received their 8 MBSR session with a trained therapist. They will be given their assignments for the week, consisting of the content of that MBSR session.
  Finally, three months after the last study session, they will be asked to return to the clinic for the follow-up assessment to complete patient-reported outcome measures.
  Arms: experimental group
Other: physiotherapy — In control group in the first session, the research program and plans for outcome assessment will be introduced. The participants then will sign the research agreement form and will be interviewed to obtain information about their pain (i.e., duration, location, and course), their medication(s), and demographics. This will be followed by the first 70-80-minute physiotherapy session. During each session, the physiotherapist will administer the Transcutaneous electrical nerve stimulation (TENS), low-level laser therapy (LLLT), and ultrasound therapy to the painful body region. In addition, they will engage in 20 minutes of exercise during each session.
  Arms: control group

SUMMARY:
It has been shown that MBSR could be effective in different types of chronic pain in geriatrics, but more evidence in the interdisciplinary context is needed.

This study is conducted to develop and compile a mindfulness-based stress reduction (MBSR) program within a context of physiotherapy rehabilitation to manage chronic pain in the elderly in an Iranian clinical setting.

The 8-session MBSR treatment protocol was translated, revised for the Iranian elderlies, and compiled as a one-on-one therapy using a unique protocol with 20-session physiotherapy. 40 volunteers aged 65 or more with musculoskeletal chronic pain will be selected and receive the program for 8 consecutive weeks with a 3-month follow-up. Treatment satisfaction levels, adherence to treatment sessions, and patient-reported clinical outcome measures were used at baseline, immediately post-intervention, and three months following the intervention, measuring pain, anxiety, fatigue, sleep disturbance, pain interference levels, and kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or more
* Have chronic pain
* Have ability of reading and writing in Persian
* Visiting the clinic in which the study was took place

Exclusion Criteria:

* Dose not have any diagnosed Cognitive Impairment
* Failure to approve the consent form

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
. The Patient Global Assessment of Treatment Satisfaction (PGATS) | At the baseline, immediately after last session, and 3-month follow-up.
  Treatment satisfaction was assessed with six questions asking the participants to rate six domains of treatment satisfaction using a 5-point Likert scale ranging from 0 ("Very dissatisfied") to 4 ("Very satisfied"). Specifically, satisfaction with the combined physiotherapy and MBSR protocol, the duration of the entire protocol, the duration of each treatment session, the content of the treatment sessions, and homework assignments were measured using this tool. Participants were also asked to rate their overall satisfaction with the treatment on the same Likert scale.
The Numerical Rating Scale-11 (NRS-11). | At the baseline, immediately after last session, and 3-month follow-up.
  Average pain intensity in the past week and post-session current pain intensity were assessed at the end of each session using the NRS-11 (0 = "no pain" and 10 = "worst pain imaginable").

SECONDARY OUTCOMES:
The Patient Reported Outcomes Measurement Information System (PROMIS-29 v2.0). | At the baseline, immediately after last session, and 3-month follow-up.
  Physical function, anxiety, depression, fatigue, sleep disturbances, ability to participate in social roles, and pain interference were assessed using the 4-item short form version of the PROMIS-29 v2.0.
The Tampa Scale Kinesiophobia (TKS-11). | At the baseline, immediately after last session, and 3-month follow-up.
  Fear of movement (i.e., kinesiophobia) was assessed using the brief (11-item) version of the TKS-1. Respondents are asked to indicate agreement with each item on a Likert scale from ("strongly disagree") to 4 ("strongly agree). The items are summed into a total score ranging from 11 to 44. Higher scores indicate a greater fear of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Reza poorhosein, PhD, Study Chair — Faculty of Psychology and Education, the University of Tehran.
Locations (1):
- Bahar physiotherapy clinic, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
Access to the results of the data starts simultaneously with the publication of an article based on them and presenting all the information in the doctoral thesis of the main researcher in 2024. The release of the raw data will be one year after the publication of the results, although the ethics committees and the doctoral thesis advising committee will have access to all the data at all stages.
Supporting Information: SAP, ICF, CSR
Time Frame: 1 year after manuscript publication.
Access Criteria: The data will be sent only to experts working in academic environments who have researches in line with the field of this study according to their request.To receive the data, one email should be send to corresponded author of this research.